CLINICAL TRIAL: NCT03619525
Title: Bedside Lung Ultrasound to Assess Lung Recruiting Maneuver With Cardiopulmonary Bypass in Valvular Cardiac Surgery.
Brief Title: Ultrasonographic Assessment of the Effect of CPB Acute Lung Injury
Acronym: CBP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maged Abdel-Wahab Abdel-Aziz, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: lung ultrasound after CPB
Record Dates: First submitted 2018-07-25; First posted 2018-08-08 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Lung Ultrasound

STUDY DESIGN:
Intervention Model Description: sixty patients aged from 18-60 years old, scheduled for elective cardiac surgery with CPB will be included in the study. Patients will be randomly allocated into one of two groups: Group A (n=30): will receive intermittent lung recruitment during CPB.Group B (n=30): control group.
Who Masked: Investigator
Masking Description: numbered, sealed opaque envelope.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- recruitment group (Active Comparator): will receive intermittent lung recruitment during CPB
  Interventions: Procedure: lung recruitment
- control group (No Intervention): will recieve no intervention

INTERVENTIONS:
Procedure: lung recruitment — During bypass, patients in this group will receive a lung protective design in the form of continuous positive airway pressure (CPAP) by closing APL valve at pressure of 5 Cm H2o combined with intermittent recruitment by sustained manual lung inflation at a pressure of 35 cmH2O for 30 seconds every (30-40) minute
  Arms: recruitment group

SUMMARY:
The study is designed to use the lung ultrasound to assess the effect of intermittent lung recruitment during cardiopulmonary bypass in cardiac surgeries on extra vascular lung water.

DETAILED DESCRIPTION:
Significant respiratory dysfunction is a common problem after cardiac surgery, with an incidence of about 25%. the formation of atelectasis appears to be the primary factor responsible for increased intrapulmonary shunt after cardiac surgery with CPB. The investigators will use the lung ultrasound to evaluate the effects of intermittent recruitment of the lungs during CPB on extra vascular lung water (EVLW).

Objectives :

To evaluate the effect of intermittent lung recruitment during CPB in cardiac surgery on:

Lung ultrasound score (LUS),Oxygenation at different times postoperatively,Time for extubation and length of ICU stay

sixty patients aged from 18-60 years old, scheduled for elective cardiac surgery with CPB will be included in the study. Patients will be randomly allocated into one of two groups: Group A (n=30): will receive intermittent lung recruitment during CPB.Group B (n=30): control group.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged (18-60 years),
* elective valvular cardiac surgery with cardiopulmonary bypass (CPB).

Exclusion Criteria:

* • Emergency surgeries.

  * coronary artery bypass graft surgery
  * patients requiring re-exploration in the immediate postoperative period (within 2hours)
  * left Ventricular ejection fraction less than 40%
  * patients with preoperative congestive heart failure, cardiogenic shock , preoperative pulmonary edema
  * pre-existing severe chronic pulmonary dysfunction (defined as pulmonary disease requiring home oxygen therapy or causing shortness of breath after 1 to 2 flights of stairs)
  * Morbid obesity
  * Renally impaired patients with creatinine more than 2 mg/dl

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-10-20 (Actual); Primary Completion 2018-11-20 (Estimated); Study Completion 2018-12-05 (Estimated)

PRIMARY OUTCOMES:
lung ultrasound score | Baseline,immediately at the end of operation. 2 hours after ICU admission
  • The change of lung ultrasound score (a score ranging fom 0/36 to 36/36 where 0/36 is best while 36/36 is worst) from the baseline values for assessment of extra vascular lung water after CBP

SECONDARY OUTCOMES:
• The value of Doppler derived E/E' ratio. | Baseline,immediately at the end of operation. 2 hours after ICU admission
• Oxygenation (po2),& (po2/fio2) | Baseline,immediately at the end of operation. 2 hours after ICU admission
  po2 is measured by mmhg units while PO2/fio2 is ratio
• Time for extubation | before extubation
Length of ICU stay | before discharge to ward up to 1 week

CONTACTS AND LOCATIONS:
Overall Officials: ahmed agaty, professor, Principal Investigator — cairro university
Locations (1):
- Cairo University, Cairo, Manil, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Volpicelli G, Mussa A, Garofalo G, Cardinale L, Casoli G, Perotto F, Fava C, Frascisco M. Bedside lung ultrasound in the assessment of alveolar-interstitial syndrome. Am J Emerg Med. 2006 Oct;24(6):689-96. doi: 10.1016/j.ajem.2006.02.013. PMID 16984837